CLINICAL TRIAL: NCT06034223
Title: Effect of Proprioceptive Training Using Head Mounted Laser in Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, Lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 0220-23
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Mechanical Neck Pain
Keywords: proprioception; joint position sense error; head mounted laser; cervical range of motion

STUDY DESIGN:
Intervention Model Description: the participants are divided into two groups, control group will recieve conventional physical therapy and experimental group will recieve proprioceptive training with conventional physcial therapy.
Who Masked: Participant
Masking Description: It is a single blinded study in which participants will be alocated in two groups using simple random sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physical Therapy + Proprioceptive Training Using Head Mounted Laser (Experimental): Conventional physical therapy along with proprioceptive training, head relocation practice that is relocating the head back to the natural head posture and to pre determined postions in range with eyes open. Tracing figure of eight with eyes open.
  3 days per week for 4 weeks, 15 repititions, 1 set.
  Interventions: Other: Proprioceptive training using head mounted laser; Other: Conventional Physical therpay
- Conventional Physical Therapy only (Other): Conventional physical therapy, cervical range of motion (flexion, extension, lateral flexion and rotation), isometric exercises of neck muscles, stretching (scalene, trapezius, sternocleidomastoid), TENS, heating pad.
  3 days per week for 4 weeks, 15 repitions, 1 set.
  Interventions: Other: Conventional Physical therpay

INTERVENTIONS:
Other: Proprioceptive training using head mounted laser — Exercises include head relocation practice, i.e., relocating the head back to the natural head posture and to pre-determined positions in range with eyes open using feedback from a laser attached to their head. And then tracing the figure of eight with the help of laser.
  Arms: Conventional Physical Therapy + Proprioceptive Training Using Head Mounted Laser
Other: Conventional Physical therpay — Conventional physical therapy for mechanical neck pain which includes cervical range of motion (flexion, extension, lateral rotation, and rotation), neck isometric exercises, stretching's (scalene, trapezius, SCM) and TENS with heating pad.

SUMMARY:
The purpose of this study is to compare the effect of conventional physical therapy with and without cervical proprioceptive training using head-mounted laser system on cervical joint position sense error, pain, cervical range of motion and neck disability index. Proprioception disturbs in any function and structural impairments that is mechanical neck pain. Different studies has been done to find out the best therapy for pain management. Aim of the researcher is to give cost-effective, not so time-consuming, most effective physical therapy treatment. A literature gap exists on the effects of proprioceptive training combined with conventional physical therapy, no studies have directly compared the effect of proprioceptive training using head-mounted laser with and without conventional physical therapy. In our clinical setting, proprioceptive training for mechanical neck pain is not used as much as it should be. It would be a new thing to add and it can be cost-effective and better treatment for symptoms resolution

DETAILED DESCRIPTION:
Mechanical neck pain (MNP) is a common condition, affecting 30% to 50% of the general population, and is most prevalent in middle age. It is responsible for reducing the quality of life and one of the leading causes of disability worldwide with annual prevalence of 48.5%. Mechanical neck pain is characterized by several structural and functional features. The causes of MNP include structural and functional impairment of cervical muscles, degenerative changes of cervical spine, arthritis, inflammation, and trauma, abnormal posture, and movements. Current studies have found that one of the main problems in patients with MNP is the impairment of cervical proprioception. decreased range of motion (ROM) and functional ability, greater muscle fatigability and a reduction in the strength and endurance capacity of the muscles.

Despite neck disorders being so common in the population, little evidence supporting effective interventions has been identified. Conservative treatments used to help manage MNP are numerous and include usual medical care various forms of exercise, massage, and acupuncture. Medications, manual therapies, and exercise are the most widely used treatment modalities for MNP. 33% of individuals with neck pain sought care from physical therapy. Physical therapy improves pain, function and patient satisfaction in adults suffering from MNP, improves neck disability index. Physical therapy treatment includes cervical and thoracic spine mobilization/manipulation techniques active and passive exercise, ultrasound, transcutaneous electrical nerve stimulation, patient education. Spinal manipulative therapy (SMT), trigger point dry needling and trigger point manual therapy.

Proprioception is the sense of perceiving self-movement, action of parts of the body and location. It is a term commonly used to describe the ascending information by the afferent receptors towards the central nervous system contributing to the neuromuscular control of movement and encompasses the sensation of joint movement (kinaesthesia) and joint position (joint position sense). Cervical spine has a very delicate proprioceptive system, which signals the position of the head relative to the trunk, coordinates the vestibular and visual systems and it plays a crucial role in controlling posture and balance and is of great importance for spatial orientation. The deficits of Proprioception of cervical spine have been associated with age, pain muscle fatigue, forward head posture, cervical spondylosis, reduced balance control and abnormal posture, decreased neck muscle strength and altered motor control in the cervical spine.

In last two decades the interest in the assessment and treatment of proprioception of the cervical spine has increased exponentially. Cervical joint position sense (JPS) is a major component of proprioception and mainly reflects the ascending input (afferent) of cervical muscle, disc, capsule, and ligament receptors. Proprioception is evaluated using the Joint Position Sense Error (JPSE), which reflects a person's ability to accurately return his head to a predefined target after a cervical movement.

Evidence to date suggests that the management of sensorimotor control disturbances due to chronic neck pain may need to address the primary causes and secondary effects of alterations in proprioceptive activity. A variety of treatments are available for cervical spine proprioception. It includes proprioception training, retraining of deep cervical flexor and extensor muscles, and etiological management of pain, strength training, cervical manipulation and acupuncture and many other conventional therapy protocols. Cervical proprioception training not only improves patient-perceived pain and disability but also has an effect on other aspects of neuromuscular function, specifically the coordination between the deep and superficial cervical flexors and balance.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age: 45 to 55 years
* Mechanical neck pain more than 3 months (chronic stage)
* Individuals having cervical radiculopathy (Spurling Test A and Spurling test B +ve)
* Decreased Range of motion (Flexion 80 to 90*) (Extension 70*) (Lateral Flexion 20 TO 45*) (Rotation 90*)
* Numeric Pain Rating Scale: 5 to 08
* Cervical spondylosis on Xray

Exclusion Criteria:

* Individuals having vascular pathology of neck.
* Previous surgery related to cervical spine.
* Individuals having structural deformity of spine (Adam's forward bend test)
* Spinal Cord Injury /Cervical Myelopathy
* Malignancy and tumor
* Infection
* Previous history of Cervical spine fractures

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
cervical joint position sense error | 4 weeks
  use to assess proprioception
bubble inclinometer | 4 weeks
  use to assess cervical range of motion
numerical pain rating scale | 4 weeks
  used for assessment of pain in which 0 means no pain and 10 means severe pain
neck disability index | 4 weeks
  used for pain related disability in which 0-4 means no disability 5-14 means mild disability 15-24 means moderate disability, 25-34 means severe disability and 35-50 means complete disability

CONTACTS AND LOCATIONS:
Overall Officials: Nida Waseem, MS-PT*, Principal Investigator — Shifa Tameer-e-millet University
Locations (1):
- Shifa Tameer-e-Millat University Islamabad, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celenay ST, Akbayrak T, Kaya DO. A Comparison of the Effects of Stabilization Exercises Plus Manual Therapy to Those of Stabilization Exercises Alone in Patients With Nonspecific Mechanical Neck Pain: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2016 Feb;46(2):44-55. doi: 10.2519/jospt.2016.5979. Epub 2016 Jan 11. PMID 26755405
- [Background] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Background] Ganesh GS, Mohanty P, Pattnaik M, Mishra C. Effectiveness of mobilization therapy and exercises in mechanical neck pain. Physiother Theory Pract. 2015 Feb;31(2):99-106. doi: 10.3109/09593985.2014.963904. Epub 2014 Sep 29. PMID 25264016
- [Background] Sarig-Bahat H. Evidence for exercise therapy in mechanical neck disorders. Man Ther. 2003 Feb;8(1):10-20. doi: 10.1054/math.2002.0480. PMID 12586557
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Background] Vincent K, Maigne JY, Fischhoff C, Lanlo O, Dagenais S. Systematic review of manual therapies for nonspecific neck pain. Joint Bone Spine. 2013 Oct;80(5):508-15. doi: 10.1016/j.jbspin.2012.10.006. Epub 2012 Nov 16. PMID 23165183
- [Background] Gross AR, Kay T, Hondras M, Goldsmith C, Haines T, Peloso P, Kennedy C, Hoving J. Manual therapy for mechanical neck disorders: a systematic review. Man Ther. 2002 Aug;7(3):131-49. doi: 10.1054/math.2002.0465. PMID 12372310
- [Background] Walker MJ, Boyles RE, Young BA, Strunce JB, Garber MB, Whitman JM, Deyle G, Wainner RS. The effectiveness of manual physical therapy and exercise for mechanical neck pain: a randomized clinical trial. Spine (Phila Pa 1976). 2008 Oct 15;33(22):2371-8. doi: 10.1097/BRS.0b013e318183391e. PMID 18923311
- [Background] Leininger B, McDonough C, Evans R, Tosteson T, Tosteson AN, Bronfort G. Cost-effectiveness of spinal manipulative therapy, supervised exercise, and home exercise for older adults with chronic neck pain. Spine J. 2016 Nov;16(11):1292-1304. doi: 10.1016/j.spinee.2016.06.014. Epub 2016 Jun 23. PMID 27345747
- [Background] Llamas-Ramos R, Pecos-Martin D, Gallego-Izquierdo T, Llamas-Ramos I, Plaza-Manzano G, Ortega-Santiago R, Cleland J, Fernandez-de-Las-Penas C. Comparison of the short-term outcomes between trigger point dry needling and trigger point manual therapy for the management of chronic mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Nov;44(11):852-61. doi: 10.2519/jospt.2014.5229. Epub 2014 Sep 30. PMID 25269764
- [Background] Strimpakos N, Sakellari V, Gioftsos G, Kapreli E, Oldham J. Cervical joint position sense: an intra- and inter-examiner reliability study. Gait Posture. 2006 Jan;23(1):22-31. doi: 10.1016/j.gaitpost.2004.11.019. PMID 16311191
- [Background] Reddy RS, Tedla JS, Dixit S, Abohashrh M. Cervical proprioception and its relationship with neck pain intensity in subjects with cervical spondylosis. BMC Musculoskelet Disord. 2019 Oct 15;20(1):447. doi: 10.1186/s12891-019-2846-z. PMID 31615495
- [Background] Reddy RS, Meziat-Filho N, Ferreira AS, Tedla JS, Kandakurti PK, Kakaraparthi VN. Comparison of neck extensor muscle endurance and cervical proprioception between asymptomatic individuals and patients with chronic neck pain. J Bodyw Mov Ther. 2021 Apr;26:180-186. doi: 10.1016/j.jbmt.2020.12.040. Epub 2020 Dec 31. PMID 33992242
- [Background] Vuillerme N, Pinsault N, Bouvier B. Cervical joint position sense is impaired in older adults. Aging Clin Exp Res. 2008 Aug;20(4):355-8. doi: 10.1007/BF03324868. PMID 18852550
- [Background] de Vries J, Ischebeck BK, Voogt LP, van der Geest JN, Janssen M, Frens MA, Kleinrensink GJ. Joint position sense error in people with neck pain: A systematic review. Man Ther. 2015 Dec;20(6):736-44. doi: 10.1016/j.math.2015.04.015. Epub 2015 May 2. PMID 25983238
- [Background] Pinsault N, Vuillerme N. Degradation of cervical joint position sense following muscular fatigue in humans. Spine (Phila Pa 1976). 2010 Feb 1;35(3):294-7. doi: 10.1097/BRS.0b013e3181b0c889. PMID 20075783
- [Background] Heikkila H, Johansson M, Wenngren BI. Effects of acupuncture, cervical manipulation and NSAID therapy on dizziness and impaired head repositioning of suspected cervical origin: a pilot study. Man Ther. 2000 Aug;5(3):151-7. doi: 10.1054/math.2000.0357. PMID 11034885
- [Background] Soysal M, Kara B, Arda MN. Assessment of physical activity in patients with chronic low back or neck pain. Turk Neurosurg. 2013;23(1):75-80. doi: 10.5137/1019-5149.JTN.6885-12.0. PMID 23344871